CLINICAL TRIAL: NCT03714763
Title: The Predictive Value of Positron Emission Tomography-Magnetic Resonance (PET-MR) Mediated Dopamine D2 Receptors Imaging in the Drug Therapy of Nonfunctioning Pituitary Adenoma
Brief Title: Dopamine D2 Receptors(D2R) Imaging in Nonfunctioning Pituitary Adenoma(NFPA)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhebao Wu (Other)
Collaborators: Xinqiao Hospital of Chongqing (Other); First Hospital of China Medical University (Other); Beijing Tiantan Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); First Affiliated Hospital of Fujian Medical University (Other); Peking Union Medical College Hospital (Other); Huashan Hospital (Other); Chinese PLA General Hospital (Other)
Responsible Party: Sponsor-Investigator, Zhebao Wu, Principal Investigator, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DD2RN-2018
Record Dates: First submitted 2018-10-14; First posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Pituitary Adenoma
Keywords: Nonfunctioning Pituitary Adenoma; Dopamine Agonist; Dopamine D2 Receptors; PET-MR
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug treatment (Experimental): Subjects who show high expression of dopamine D2 receptors in PET-MR imaging.
  Interventions: Drug: Drug treatment
- Surgery (Experimental): Subjects who show low expression of dopamine D2 receptors in PET-MR imaging.
  Interventions: Other: Surgery

INTERVENTIONS:
Drug: Drug treatment — Subjects who show high expression of dopamine D2 receptors in PET-MR imaging will be treated with Cabergoline(CAB) tablets 2mg/week or bromocriptine(BC) tablets 7.5mg/ day.The pituitary hormone levels, tumor volume, visual acuity and visual field scale will be measured every 3 months. The medication will be stopped if failure to decrease tumor size and the subjects will be advised to surgical therapy.
  Arms: Drug treatment
Other: Surgery — Subjects who show low expression of dopamine D2 receptors in PET-MR imaging will be treated with endoscopic transphenoidal pituitary surgery .
  Arms: Surgery

SUMMARY:
To study the in vivo expression of dopamine D2 receptors in nonfunctioning pituitary adenoma and the predictive role of dopamine dopamine D2 receptors PET-MR imaging in the therapeutic effect of dopamine agonists（DA）.

DETAILED DESCRIPTION:
Dopamine agonists are the first line therapy for prolactinoma,which are also effective in some cases of other subtypes of pituitary tumors. It had been showed that dopamine agonists inhibit prolactin secretion by binding to and activating dopamine D2 receptors. PET-MR combined MR images with PET function images is substantial to evaluate the expression of dopamine D2 receptors.The aim is to study the in vivo expression of dopamine D2 receptors in prolactinoma and the predictive role of dopamine D2 receptors PET-MR imaging in the therapeutic effect of dopamine agonists.

ELIGIBILITY:
Inclusion Criteria:

1. Normal serum pituitary hormone levels or mild increase of serum prolactin.
2. Enhanced MRI shows a pituitary tumor and tumor diameter>1cm.
3. Aged between 18 and 65 years old, either sex.
4. Karnofsky performance status ≥ 70.
5. The patient has signed the informed consent.

Exclusion Criteria:

1. Patients concomitantly taking the psychotropic drugs.
2. Patients with parkinson disease and is taking dopaminergic agents.
3. Patients with pituitary adenoma who received Gamma knife treatment.
4. Pregnant or lactating women.
5. Patients with poor compliance, who cannot implement the program strictly.
6. History of allergic reactions attributed to compounds of similar chemical or biologic composition to cabergoline.
7. Patients with claustrophobia. -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on tumor volume | Up to 6 months]
  Change from baseline on tumor volume measured by enhanced pituitary Magnetic Resonance Imaging（MRI）.
  Record the tumor volume from enhanced pituitary MRI on every 3 month follow-up visit.

SECONDARY OUTCOMES:
Change from baseline of visual acuity | Up to 6 months
  Record the Visual acuity on every 3 month follow-up visit.
Change from visual field scale | Up to 6 months
  2.Record the Visual field scale on every 3 month follow-up visit, 0 = normal, no vision loss; 1 = one quadrant vision loss; 2 = two quadrants of vision loss; 3 = three quadrants of vision loss; 4 = four quadrants of vision loss but retain a central tubular vision; 5 = blind

IPD SHARING:
Plan to Share IPD: No
The individual patient Data would not be shared to the third facility, but the sponsor hasn't decided whether to share the individual patient date to the other related studies hold by himself in the future.

REFERENCES:
- [Result] Mukherjee J, Majji D, Kaur J, Constantinescu CC, Narayanan TK, Shi B, Nour MT, Pan ML. PET radiotracer development for imaging high-affinity state of dopamine D2 and D3 receptors: Binding studies of fluorine-18 labeled aminotetralins in rodents. Synapse. 2017 Mar;71(3):10.1002/syn.21950. doi: 10.1002/syn.21950. Epub 2016 Nov 30. PMID 27864853
- [Result] Cooper O, Melmed S. Subclinical hyperfunctioning pituitary adenomas: the silent tumors. Best Pract Res Clin Endocrinol Metab. 2012 Aug;26(4):447-60. doi: 10.1016/j.beem.2012.01.002. Epub 2012 May 22. PMID 22863387
- [Result] Colao A, Di Somma C, Pivonello R, Faggiano A, Lombardi G, Savastano S. Medical therapy for clinically non-functioning pituitary adenomas. Endocr Relat Cancer. 2008 Dec;15(4):905-15. doi: 10.1677/ERC-08-0181. Epub 2008 Sep 9. PMID 18780796
- [Result] Su Z, Wang C, Wu J, Jiang X, Chen Y, Chen Y, Zheng W, Zhuge Q, Wu Z, Zeng Y. Expression of dopamine 2 receptor subtype mRNA in clinically nonfunctioning pituitary adenomas. Neurol Sci. 2012 Apr;33(2):275-9. doi: 10.1007/s10072-011-0701-6. Epub 2011 Jul 12. PMID 21748460